CLINICAL TRIAL: NCT03095638
Title: A 2-Part, Phase I, Single Dose, Crossover Relative Bioavailability Study of Both TIVICAY 10 mg Conventional Tablets and 5 mg Dispersible Tablets Compared to Conventional TIVICAY Tablets in Fasted Healthy Adult Subjects
Brief Title: Bioavailability Study of 10 Milligram (mg) and 5 mg Tablets Versus Conventional Tablets of Dolutegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205893
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2018-12-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
Keywords: Dispersible tablets; Bioavailability; Dolutegravir; Healthy; Conventional tablets
MeSH Terms: conditions — HIV Infections | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Treatment sequence A/B: Part 1 (Experimental): Eligible subjects will be randomized in sequence A/B in Part 1 and will receive A: conventional 10 mg DTG tablet (5 tablets) in Period 1 and B: conventional 50 mg DTG tablet in Period 2, administered directly to mouth.
  Interventions: Drug: Conventional dolutegravir 10 mg tablet; Drug: Conventional dolutegravir 50 mg tablet
- Treatment sequence B/A: Part 1 (Experimental): Eligible subjects will be randomized in sequence B/A in Part 1 and will receive B: conventional 50 mg DTG tablet in Period 1 and A: conventional 10 mg DTG tablet (5 tablets) in Period 2, administered directly to mouth.
  Interventions: Drug: Conventional dolutegravir 10 mg tablet; Drug: Conventional dolutegravir 50 mg tablet
- Treatment sequence C/D/E: Part 2 (Experimental): Eligible subjects will be randomized in sequence C/D/E in Part 2 and will receive C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 1, D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 2 and E: conventional 25 mg DTG tablet administered as direct to mouth in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet
- Treatment sequence D/E/C: Part 2 (Experimental): Eligible subjects will be randomized in sequence D/E/C in Part 2 and will receive D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 1, E: conventional 25 mg DTG tablet administered as direct to mouth in Period 2 and C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet
- Treatment sequence E/C/D: Part 2 (Experimental): Eligible subjects will be randomized in sequence E/C/D in Part 2 and will receive E: conventional 25 mg DTG tablet administered as direct to mouth in Period 1, C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 2 and D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet
- Treatment sequence C/E/D: Part 2 (Experimental): Eligible subjects will be randomized in sequence C/E/D in Part 2 and will receive C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 1, E: conventional 25 mg DTG tablet administered as direct to mouth in Period 2 and D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet
- Treatment sequence D/C/E: Part 2 (Experimental): Eligible subjects will be randomized in sequence D/C/E in Part 2 and will receive D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 1, C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 2 and E: conventional 25 mg DTG tablet administered as direct to mouth in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet
- Treatment sequence E/D/C: Part 2 (Experimental): Eligible subjects will be randomized in sequence E/D/C in Part 2 and will receive E: conventional 25 mg DTG tablet administered as direct to mouth in Period 1, D: 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth in Period 2 and C: 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken in Period 3.
  Interventions: Drug: Dispersible dolutegravir 5 mg tablet; Drug: Conventional dolutegravir 25 mg tablet

INTERVENTIONS:
Drug: Conventional dolutegravir 10 mg tablet — Single dose of five 10 mg DTG tablets will be administered directly to mouth with 240 mL of water in the morning to randomized subjects in fasting state present in Part 1. DTG will be a white, round shaped, biconvex tablet.
  Arms: Treatment sequence A/B: Part 1; Treatment sequence B/A: Part 1
Drug: Conventional dolutegravir 50 mg tablet — Single dose of one 50 mg tablet will be administered directly to mouth with 240 mL of water in the morning to randomized subjects in fasting state present in Part 1. DTG will be a white, round shaped, biconvex tablet.
  Arms: Treatment sequence A/B: Part 1; Treatment sequence B/A: Part 1
Drug: Dispersible dolutegravir 5 mg tablet — Single dose of five 5 mg DTG tablets will be administered as dispersed in water or direct to mouth with 240 mL of water in the morning to randomized subjects in fasting state present in Part 2. DTG will be a white, round shaped, biconvex tablet.
  Arms: Treatment sequence C/D/E: Part 2; Treatment sequence C/E/D: Part 2; Treatment sequence D/C/E: Part 2; Treatment sequence D/E/C: Part 2; Treatment sequence E/C/D: Part 2; Treatment sequence E/D/C: Part 2
Drug: Conventional dolutegravir 25 mg tablet — Single dose of one 25 mg DTG tablet will be administered directly to mouth with 240 mL of water in the morning to randomized subjects in fasting state present in Part 2. DTG will be a white, round shaped, biconvex tablet.
  Arms: Treatment sequence C/D/E: Part 2; Treatment sequence C/E/D: Part 2; Treatment sequence D/C/E: Part 2; Treatment sequence D/E/C: Part 2; Treatment sequence E/C/D: Part 2; Treatment sequence E/D/C: Part 2

SUMMARY:
The aim of this cross-over study is to compare the relative bioavailability and pharmacokinetic parameters of both 10 mg conventional tablets and 5 mg dispersible tablets of dolutegravir (DTG) with that of 25 mg or 50 mg conventional DTG tablets. The study will be carried out in 2 parts. Part 1 of the study will be open-label, 2 period designs with a wash out period of at least 7 days between the dosing periods. Subjects will be randomized to receive either single dose of five 10 mg DTG tablets or one 50 mg DTG tablet in a crossover manner in the fasting state. Part 2 of the study will be a 3 period crossover design with a wash out period of at least 7 days between the dosing periods. Subjects will be randomized to receive either single dose of five 5 mg DTG tablets (administered as dispersed with water or directly to mouth) or one 25 mg DTG tablet in a crossover manner in the fasting state. Subjects will have a follow-up visit 7-10 days post last dose of study treatment. Approximately 14 healthy subjects will participate in Part 1 and approximately 24 healthy subjects will participate in Part 2 of the study. The total duration of Part 1 will be approximately 7 to 8 weeks and that of part 2 will be approximately 8 to 9 weeks.

TIVICAY® is a trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history and electrocardiogram [ECG]). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) for males and >= 45 kg for females and body mass index (BMI) within the range 18.5 - 31.0 kg per meter square (kg/m^2) (inclusive).
* Male or female. Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 2 weeks after dosing with study medication and completion of the follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Alanine amino transferase (ALT) and bilirubin >1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT correction using Fridericia Formula (QTcF) >450 Milliseconds (msec).
* Unable to refrain from the use of prescription [that is (i.e. or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine- containing products within 1 month prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Creatinine clearance (CrCL) <90 mL/minute.
* A positive hepatitis B surface antigen (HBsAg) or a positive hepatitis B core antibody with a negative hepatitis B surface antibody, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immuno-deficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Derived] Singh RP, Adkison KK, Baker M, Parasrampuria R, Wolstenholme A, Davies M, Sewell N, Brothers C, Buchanan AM. Development of Dolutegravir Single-entity and Fixed-dose Combination Formulations for Children. Pediatr Infect Dis J. 2022 Mar 1;41(3):230-237. doi: 10.1097/INF.0000000000003366. PMID 34817414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 site in the United States of America from 03 May 2017 to 23 Jun 2017. The study was conducted in 2 parts and a total of 38 participants were enrolled: 14 in Part 1 (treatment A and B over 2 dosing periods) and 24 in Part 2 (treatment C,D,E, over 3 dosing periods) with washout of 7(-4 hours) days between doses.
Pre-assignment Details: A total of 106 participants were screened however 68 were screen failures the reasons for which were did not meet inclusion/exclusion, adverse event, lost to follow up, investigator discretion, withdrew consent and screened but enrollment target reached prior to enrollment. All of the 38 enrolled participants completed the study.
Groups:
- DTG 10 mg Followed by DTG 50 mg: Part 1: Participants in Part 1 (P1), received Five 10 milligrams (mg) Dolutegravir [DTG] tablets direct to mouth with 240 milliliters (mL) of water in Treatment Period 1 followed by One 50 mg DTG tablet direct to mouth with 240 mL of water in Treatment Period 2. There was a washout of 7(-4 hours) days between the treatment periods 1 and 2.
- DTG 50 mg Followed by DTG 10 mg: Part 1: Participants in P1, received One 50 mg DTG tablet direct to mouth with 240 mL of water in Treatment Period 1 followed by Five 10 mg DTG tablets direct to mouth with 240 mL of water in Treatment Period 2. There was a washout of 7(-4 hours) days between the treatment periods 1 and 2.
- DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2: Participants in P2, received Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in Treatment Period 1, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 2) in Treatment Period 2, followed by Conventional 25 mg DTG tablet administered as direct to mouth [reference]) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2: Participants in P2, received Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 2) in Treatment Period 1, followed by Conventional 25 mg DTG tablet administered as direct to mouth (reference) in Treatment Period 2, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2: Participants in P2, received Conventional 25 mg DTG tablet administered as direct to mouth (reference) in Treatment Period 1, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in Treatment Period 2, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 2) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2: Participants in P2, received Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in Treatment Period 1, followed by Conventional 25 mg DTG tablet administered as direct to mouth (reference) in Treatment Period 2, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 2) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2: Participants in P2, received Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 2) in Treatment Period 1, followed by (Dispersible 5 mg DTG tablet [5 tablets] administered as a dispersion and immediately taken (test 1) in Treatment Period 2, followed by Conventional 25 mg DTG tablet administered as direct to mouth (reference) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2: Participants in P2, received Conventional 25 mg DTG tablet administered as direct to mouth (reference) in Treatment Period 1, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 2) in Treatment Period 2, followed by Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in Treatment Period 3. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
Period: P1: Period 1 (4 Days)
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P1: Period 1, Washout (7 [-4 Hours])
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P1: Period 2 (4 Days)
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P1: Period 2, Washout (7[-4 Hours])
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 1 (4 Days)
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 1, Washout (7[-4 Hours])
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 2 (4 Days)
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 2, Washout (7[-4 Hours])
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 3 (4 Days)
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2: Period 3, Washout (7[-4 Hours])
Arm/Group | DTG 10 mg Followed by DTG 50 mg: Part 1 | DTG 50 mg Followed by DTG 10 mg: Part 1 | DTG 5 mg (Test 1) Then DTG 5 mg (Test 2) Then by DTG 25 mg: P2 | DTG 5 mg Then DTG 25 mg (Reference) Then DTG 5 mg: Part 2 | DTG 25 mg (Reference) DTG 5 mg Followed by DTG 5 mg: P2 | DTG 5 mg Then DTG 25 mg Then DTG 5 mg: P2 | DTG 5 mg Followed by DTG 5 mg Followed by DTG 25 mg: Part 2 | DTG 25 mg Followed by DTG 5 mg Followed by DTG 5 mg: Part 2
Started | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Participants: Part 1: Participants in Part 1 of the study received each of 2 treatments Five 10 mg DTG tablets direct to mouth with 240 mL of water and One 50 mg DTG tablet direct to mouth with 240 mL of water over 2 Treatment periods. There was a washout of at least 7 (-4 hours) days between the Treatment Periods 1 and 2.
- Total Participants: Part 2: Participants in Part 2, of the study received each of the 3 treatments Dispersible 5 mg DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1), Dispersible 5 mg DTG tablet (5 tablets) administered as direct to mouth (test 1) and Conventional 25-mg DTG tablet administered as direct to mouth [reference]) over 3 Treatment Periods. There was a washout of 7(-4 hours) days between the treatment periods 1, 2 and 3.
- Total: Total of all reporting groups
Arm/Group | Total Participants: Part 1 | Total Participants: Part 2 | Total
Number analyzed (Participants) | 14 | 24 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (9.00) | 35.7 (9.71) | 34.9 (9.355)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 5 | 16 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 9 | 13
  White | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Dose Extrapolated to Infinite Time (AUC[0-infinity]) of DTG for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the pharmacokinetic (PK) profile of DTG tablets in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times. The PK Population was defined as participants in the All Subjects Population for whom a PK sample was obtained and that had evaluable PK assay results.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/mL (h*ng/mL)
Groups:
- DTG 10 mg: Participants in this cross-over study received 10 mg DTG tablet (5 tablets) administered direct to mouth (test) in either of the 2 dosing periods in Part 1 as per randomization schedule. Both the dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- DTG 50 mg: Participants in this cross-over study received 50 mg DTG tablet administered direct to mouth (reference) in either of the 2 dosing periods in Part 1 as per randomization schedule. Both the dosing periods were separated by a washout of 7(-4 hours) days between the doses.
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
hours*nanograms/mL (h*ng/mL) | 58900 (37.2) | 58400 (29.3)
Statistical Analysis 1: Comparison: DTG 10 mg vs DTG 50 mg; Test type: Other; Ratio = 1.0084, 90% CI 2-sided [0.8626 to 1.1789]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Dose to Last Measurable Concentration AUC [0-t] of DTG for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the PK profile of DTG tablets in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times..
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
h*ng/mL | 55800 (36.6) | 55200 (27.3)
Statistical Analysis 1: Comparison: DTG 10 mg vs DTG 50 mg; Test type: Other; Ratio = 1.0121, 90% CI 2-sided [0.8648 to 1.1845]

3. Primary Outcome: Maximum Observed Concentration (Cmax) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
nanograms/milliliter (ng/mL) | 2780 (42.1) | 2700 (25.7)
Statistical Analysis 1: Comparison: DTG 10 mg vs DTG 50 mg; Test type: Other; Ration = 1.0329, 90% CI 2-sided [0.8623 to 1.2373]

4. Primary Outcome: AUC (0-infinity) of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- DTG 5 mg (Test 1): Participants in this cross-over study received 5 mg dispersible DTG tablet (5 tablets) administered as a dispersion and immediately taken (test 1) in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- DTG 5 mg (Test 2): Participants in this cross-over study received 5 mg dispersible DTG tablet (5 tablets) administered as direct to mouth (test 2) in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- DTG 25 mg (Reference): Participants in this cross-over study received 25 mg DTG tablet administered as direct to mouth (reference) in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
h*ng/mL | 51300 (18.8) | 48800 (26.9) | 31600 (34.4)
Statistical Analysis 1: Comparison: DTG 5 mg (Test 1) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.6242, 90% CI 2-sided [1.4986 to 1.7604]
Statistical Analysis 2: Comparison: DTG 5 mg (Test 2) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.5448, 90% CI 2-sided [1.4253 to 1.6743]

5. Secondary Outcome: AUC (0-t) of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
h*ng/mL | 49000 (17.5) | 46700 (26.0) | 30100 (33.7)
Statistical Analysis 1: Comparison: DTG 5 mg (Test 1) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.6292, 90% CI 2-sided [1.5030 to 1.7661]
Statistical Analysis 2: Comparison: DTG 5 mg (Test 2) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.5519, 90% CI 2-sided [1.4317 to 1.6822]

6. Secondary Outcome: Cmax of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 2690 (24.2) | 2700 (31.5) | 1500 (34.2)
Statistical Analysis 1: Comparison: DTG 5 mg (Test 1) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.7933, 90% CI 2-sided [1.6226 to 1.9819]
Statistical Analysis 2: Comparison: DTG 5 mg (Test 2) vs DTG 25 mg (Reference); Test type: Other; Ratio = 1.7974, 90% CI 2-sided [1.6263 to 1.9865]

7. Secondary Outcome: Plasma DTG Lag Time Before Observation of Drug Concentrations (Tlag) for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

8. Secondary Outcome: Time to First Occurrence of Cmax (Tmax) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
hours | 2.01 [1.00 to 6.00] | 2.00 [0.50 to 5.03]

9. Secondary Outcome: Terminal Phase Half-life (t1/2) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
hours | 15.81 (22.7) | 16.23 (20.8)

10. Secondary Outcome: Terminal-phase Rate Constant (Lambda z) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
per hour | 0.0439 (22.7) | 0.0427 (20.8)

11. Secondary Outcome: Percentage of AUC (0-infinity) Obtained by Extrapolation (%AUCex) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Mean (95% Confidence Interval); unit: Percentage of AUC
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Percentage of AUC | 5.17 [2.96 to 7.38] | 5.52 [3.43 to 7.61]

12. Secondary Outcome: Area Under the Concentration-time Curve Over Time Zero (Pre-dose) to 24 Hours After Dose Administration (AUC[0-24]) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
h*ng/mL | 37500 (38.1) | 36600 (24.3)

13. Secondary Outcome: Apparent Oral Clearance (CL/F) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Liters/hour | 0.849 (37.2) | 0.856 (29.3)

14. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- DTG 50 mg: Participants in this cross-over study received treatment B in either of the 2 dosing periods in Part 1 as per randomization schedule. Both the dosing periods were separated by a washout of 7(-4 hours) days between the doses.
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Liters | 19.4 (39.2) | 20.0 (22.8)

15. Secondary Outcome: Last Observed Quantifiable Concentration (Ct) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
ng/mL | 106 (72.8) | 114 (73.5)

16. Secondary Outcome: Observed Concentration at 24 Hours After Dose Administration (C24) of DTG for Part 1
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
ng/mL | 912 (37.2) | 916 (29.4)

17. Secondary Outcome: Plasma DTG Tlag for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

18. Secondary Outcome: Tmax of DTG for Part 2
Description: Blood sample were collected at the indicated time points after administration of study treatment to investigate the pharmacokinetic profile of DTG tablets in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
hours | 1.00 [0.50 to 6.00] | 1.00 [0.50 to 5.00] | 1.75 [0.50 to 4.00]

19. Secondary Outcome: t1/2 of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
hours | 15.66 (15.3) | 15.48 (14.3) | 15.78 (14.7)

20. Secondary Outcome: Lambda Z of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
per hour | 0.0443 (15.3) | 0.0448 (14.3) | 0.0439 (14.7)

21. Secondary Outcome: %AUCex of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Mean (95% Confidence Interval); unit: Percentage of AUC
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Percentage of AUC | 4.37 [3.39 to 5.35] | 4.23 [3.35 to 5.11] | 4.66 [3.61 to 5.71]

22. Secondary Outcome: AUC (0-24) of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
h*ng/mL | 34000 (16.1) | 32300 (24.9) | 20400 (32.7)

23. Secondary Outcome: DTG CL/F for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Groups:
- DTG 5 mg (Test 1): Participants in this cross-over study received treatment C in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- DTG 5 mg (Test 2): Participants in this cross-over study received treatment D in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- DTG 25 mg (Reference): Participants in this cross-over study received treatment E in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Liters/hour | 0.487 (18.8) | 0.513 (26.9) | 0.792 (34.4)

24. Secondary Outcome: Vz/F of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Liters | 11.0 (15.8) | 11.4 (24.6) | 18.0 (33.5)

25. Secondary Outcome: Ct of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 89.3 (45.7) | 84.4 (48.0) | 58.2 (54.7)

26. Secondary Outcome: C24 of DTG for Part 2
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 770 (19.0) | 741 (26.9) | 493 (36.0)

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) for Part 1
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Data has been presented for AEs and SAEs up-to follow-up (25 days) in Part 1. All Subjects Population was defined as all participants who received at least 1 dose of study medication.
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Participants
  Any AE | 1 | 2
  Any SAE | 0 | 0

28. Secondary Outcome: Number of Participants With Adverse Events AEs and Serious Adverse Events SAEs for Part 2
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Data has been presented for AEs and SAEs up-to follow-up (36 days) in Part 2.
Time Frame: Up to 36 days in Part 2
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Any AE | 2 | 2 | 3
  Any SAE | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters Serum Glucose, Serum Calcium, Serum Potassium, Serum Sodium, Serum Urea for Part 1
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum glucose, serum calcium, serum potassium, serum sodium, serum urea results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: millimoles/liter (mmol/L)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
millimoles/liter (mmol/L)
  Serum glucose, Day 2, n=14, 14 | -0.091 (0.2796) | 0.071 (0.2641)
  Serum glucose, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum glucose, Follow-up, n=5, 5 | -0.178 (0.5554) | 0.022 (0.4315)
  Serum calcium, Day 2, n=14, 14 | 0.001 (0.0679) | -0.005 (0.0682)
  Serum calcium, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum calcium, Follow-up, n=5, 5 | -0.024 (0.0764) | -0.044 (0.0537)
  Serum Potassium, Day 2, n=14, 14 | 0.08 (0.258) | 0.09 (0.300)
  Serum Potassium, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Potassium, Follow-up, n=5, 5 | -0.26 (0.182) | -0.26 (0.207)
  Serum Sodium, Day 2, n=14, 14 | -1.3 (2.20) | -0.7 (2.23)
  Serum Sodium, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Sodium, Follow-up, n=5, 5 | -1.6 (1.14) | -0.6 (1.82)
  Serum Urea, Day 2, n=14, 14 | -0.394 (1.2216) | -0.444 (1.1499)
  Serum Urea, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Urea, Follow-up, n=5, 5 | 0.248 (1.6064) | -0.248 (1.6173)

30. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Alanine Amino Transferase (ALT), Serum Alkaline Phosphatase, Serum Aspartate Amino Transferase (AST), Serum Creatine Kinase for Part 1
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum ALT, serum alkaline phosphatase, serum AST, serum creatine kinase results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: International units/liter (IU/L)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
International units/liter (IU/L)
  Serum ALT, Day 2, n=14, 14 | 0.8 (6.29) | -1.1 (2.18)
  Serum ALT, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum ALT, Follow-up, n=5, 5 | -1.6 (3.58) | -1.0 (2.00)
  Serum alkaline phosphatase, Day 2, n=14, 14 | 1.5 (3.98) | 0.8 (3.12)
  Serum alkaline phosphatase, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum alkaline phosphatase, Follow-up, n=5, 5 | 1.4 (2.19) | 1.0 (5.00)
  Serum AST, Day 2, n=14, 14 | 0.6 (4.88) | -0.9 (1.29)
  Serum AST, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum AST, Follow-up, n=5, 5 | -1.0 (3.32) | 0.6 (0.89)
  Serum creatine kinase, Day 2, n=14, 14 | -43.6 (64.32) | -37.1 (52.19)
  Serum creatine kinase, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum creatine kinase, Follow-up, n=5, 5 | -17.2 (33.21) | 0.8 (22.75)

31. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 1
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum albumin and serum protein results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Grams/liter (g/L)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Grams/liter (g/L)
  Serum Albumin, Day 2, n=14, 14 | 0.3 (1.94) | 0.1 (1.79)
  Serum Albumin, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Albumin, Follow-up, n=5, 5 | -1.2 (1.30) | -0.4 (1.82)
  Serum Protein, Day 2, n=14, 14 | 2.3 (3.83) | 2.4 (3.76)
  Serum Protein, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Protein, Follow-up, n=5, 5 | 0.8 (1.79) | 1.8 (3.27)

32. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin, Serum Creatinine and Serum Direct Bilirubin for Part 1
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum bilirubin, serum creatinine and serum direct bilirubin results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: micromoles/liter (umol/L)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
micromoles/liter (umol/L)
  Serum Bilirubin, Day 2, n=14, 14 | 3.29 (3.673) | 3.28 (3.005)
  Serum Bilirubin, Follow-u, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Bilirubin, Follow-u, n=5, 5 | 0.10 (0.977) | 2.16 (3.109)
  Serum Creatinine, Day 2, n=14, 14 | 9.91 (5.791) | 11.19 (3.522)
  Serum Creatinine, Follow-u, n=5, 5: number analyzed (Participants) | 5 | 5
  Serum Creatinine, Follow-u, n=5, 5 | 4.58 (4.289) | 3.18 (4.164)
  Serum direct bilirubin, Day 2, n=14, 14 | 0.24 (0.503) | 0.30 (0.342)
  Serum direct bilirubin, Follow-up, n=5,5: number analyzed (Participants) | 5 | 5
  Serum direct bilirubin, Follow-up, n=5,5 | 0.10 (0.141) | 0.44 (0.428)

33. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Glucose, Serum Calcium, Serum Potassium, Serum Sodium, Serum Urea for Part 2
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum glucose, serum calcium, serum potassium, serum sodium, serum urea results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
mmol/L
  Serum Glucose, Day 2, n=24, 24, 24 | -0.220 (0.3653) | -0.223 (0.2715) | -0.187 (0.3599)
  Serum Glucose, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Glucose, Follow-up, n=3, 2, 3 | 0.130 (0.2506) | -0.060 (0.1556) | -0.150 (0.1559)
  Serum Calcium, Day 2, n=24, 24, 24 | 0.008 (0.0908) | 0.056 (0.0901) | 0.036 (0.0827)
  Serum Calcium, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Calcium, Follow-up, n=3, 2, 3 | 0.087 (0.0603) | -0.035 (0.0919) | -0.010 (0.0529)
  Serum Potassium, Day 2, n=24, 24, 24 | 0.00 (0.277) | 0.04 (0.298) | 0.19 (0.292)
  Serum Potassium, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Potassium, Follow-up, n=3, 2, 3 | -0.03 (0.208) | 0.05 (0.212) | -0.27 (0.208)
  Serum Sodium, Day 2, n=24, 24, 24 | -0.3 (2.37) | 0.2 (2.02) | -0.4 (2.62)
  Serum Sodium, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Sodium, Follow-up, n=3, 2, 3 | 1.3 (2.89) | 0.5 (0.71) | 0.0 (3.46)
  Serum Urea, Day 2, n=24, 24, 24 | -0.868 (1.3581) | -0.366 (0.8349) | -0.376 (1.1319)
  Serum Urea, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Urea, Follow-up, n=3, 2, 3 | 0.067 (1.5150) | -0.585 (1.2374) | -1.237 (0.6561)

34. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum ALT, Serum Alkaline Phosphate, Serum AST, Serum Creatine Kinase for Part 2
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum ALT, serum alkaline phosphatase, serum AST, serum creatine kinase results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
IU/L
  Serum ALT, Day 2, n=24, 24, 24 | -0.4 (1.72) | -1.0 (2.07) | -1.1 (1.57)
  Serum ALT, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum ALT, Follow-up, n=3, 2, 3 | 2.0 (1.73) | -1.0 (1.41) | 0.3 (2.08)
  Serum alkaline phosphatase, Day 2, n=24, 24, 24 | 0.5 (3.39) | 1.8 (3.98) | 0.2 (5.10)
  Serum alkaline phosphatase, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum alkaline phosphatase, Follow-up, n=3, 2, 3 | 4.3 (2.52) | 1.0 (11.31) | 2.3 (3.51)
  Serum AST, Day 2, n=24, 24, 24 | -1.4 (2.72) | -0.7 (1.99) | -1.3 (1.66)
  Serum AST, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum AST, Follow-up, n=3, 2, 3 | 0.0 (1.00) | -3.0 (1.41) | -0.3 (3.21)
  Serum Creatine kinase, Day 2, n=24, 24, 24 | -35.2 (67.19) | -15.7 (37.79) | -37.2 (42.81)
  Serum Creatine kinase, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Creatine kinase, Follow-up, n=3, 2, 3 | -7.3 (18.04) | -10.5 (9.19) | 23.3 (43.25)

35. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 2
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum albumin and serum protein results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
g/L
  Serum Albumin, Day 2, n=24, 24, 24 | 0.4 (2.22) | 1.1 (2.24) | 0.5 (2.47)
  Serum Albumin, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Albumin, Follow-up, n=3, 2, 3 | 2.0 (1.73) | -1.0 (4.24) | 1.7 (0.58)
  Serum Protein, Day 2, n=24, 24, 24 | 2.3 (3.29) | 3.2 (3.48) | 2.7 (3.83)
  Serum Protein, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Protein, Follow-up, n=3, 2, 3 | 1.7 (3.06) | -4.0 (7.07) | 0.3 (1.15)

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin, Serum Creatine and Serum Direct Bilirubin for Part 2
Description: Blood samples for the assessment of chemistry parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for serum bilirubin, serum creatine and serum direct bilirubin results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
umol/L
  Serum Bilirubin, Day 2, n=24, 24, 24 | 2.26 (2.26) | 2.85 (2.140) | 2.91 (2.835)
  Serum Bilirubin, Follow-u, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Bilirubin, Follow-u, n=3, 2, 3 | 0.97 (1.553) | -0.80 (1.414) | 3.07 (3.612)
  Serum Creatinine, Day 2, n=24, 24, 24 | 8.02 (4.817) | 9.83 (4.184) | 8.31 (4.218)
  Serum Creatinine, Follow-u, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum Creatinine, Follow-u, n=3, 2, 3 | 2.33 (3.293) | -4.80 (1.838) | -5.00 (6.539)
  Serum direct bilirubin, Day 2, n=24, 24, 24 | 0.33 (0.464) | 0.26 (0.388) | 0.36 (0.526)
  Serum direct bilirubin, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Serum direct bilirubin, Follow-up, n=3, 2, 3 | -0.07 (0.153) | -0.45 (0.354) | 0.30 (0.529)

37. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocyte Mean Corpuscular Hemoglobin (MCH) for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocyte MCH results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Picograms (pg)
  Blood erythrocyte MCH, Day 2, n=14, 14 | 0.08 (0.426) | -0.02 (0.283)
  Blood erythrocyte MCH, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood erythrocyte MCH, Follow-up, n=5, 5 | 0.00 (0.292) | -0.22 (0.286)

38. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocyte Mean Corpuscular Volume (MCV) for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocyte MCV results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Femtoliters (fL)
  Blood erythrocyte MCV, Day 2, n=14, 14 | -0.01 (0.598) | 0.26 (0.418)
  Blood erythrocyte MCV, Follow-up, n=5,5: number analyzed (Participants) | 5 | 5
  Blood erythrocyte MCV, Follow-up, n=5,5 | -0.38 (0.277) | 0.26 (0.416)

39. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils, Blood Platelets for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils, blood platelets results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles)
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
10^9 cells/Liter
  Blood basophils, Day 2, n=14, 14 | -0.004 (0.0101) | -0.013 (0.0230)
  Blood basophils, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood basophils, Follow-up, n=5, 5 | -0.004 (0.0195) | -0.004 (0.0230)
  Blood eosinophils, Day 2, n=14, 14 | 0.003 (0.0324) | -0.014 (0.0527)
  Blood eosinophils, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood eosinophils, Follow-up, n=5, 5 | -0.002 (0.0164) | -0.072 (0.1666)
  Blood leukocytes, Day 2, n=14, 14 | -0.33 (0.574) | -0.54 (0.633)
  Blood leukocytes, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood leukocytes, Follow-up, n=5, 5 | -0.06 (0.853) | -0.26 (0.631)
  Blood lymphocytes, Day 2, n=14, 14 | 0.018 (0.2404) | 0.049 (0.5629)
  Blood lymphocytes, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood lymphocytes, Follow-up, n=5, 5 | 0.022 (0.1894) | 0.130 (0.4077)
  Blood monocytes, Day 2, n=14, 14 | -0.031 (0.0611) | -0.064 (0.0773)
  Blood monocytes, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood monocytes, Follow-up, n=5, 5 | -0.036 (0.0740) | -0.040 (0.1279)
  Blood neutrophils, Day 2, n=14, 14 | -0.317 (0.3704) | -0.486 (0.4733)
  Blood neutrophils, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood neutrophils, Follow-up, n=5, 5 | -0.062 (0.6518) | -0.264 (0.3824)
  Blood platelets, Day 2, n=14, 14 | 14.0 (15.56) | 12.6 (18.21)
  Blood platelets, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood platelets, Follow-up, n=5, 5 | -11.2 (11.12) | 11.0 (29.56)

40. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hemoglobin for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood hemoglobin results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles)
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
g/L
  Blood hemoglobin, Day 2, n=14, 14 | 4.9 (4.36) | 4.0 (5.14)
  Blood hemoglobin, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood hemoglobin, Follow-up, n=5, 5 | -0.8 (5.50) | -3.4 (5.98)

41. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood hematocrit results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Proportion of red blood cells in blood
  Blood hematocrit, Day 2, n=14, 14 | 0.0137 (0.01585) | 0.0131 (0.01353)
  Blood hematocrit, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood hematocrit, Follow-up, n=5, 5 | -0.0042 (0.01462) | -0.0058 (0.01878)

42. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocytes for Part 1
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 25) in Part 1. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocyte results for Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles).
Time Frame: Baseline and up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
10^12 cells/Liter
  Blood erythrocytes, Day 2, n=14, 14 | 0.182 (0.1679) | 0.193 (0.1616)
  Blood erythrocyte, Follow-up, n=5, 5: number analyzed (Participants) | 5 | 5
  Blood erythrocyte, Follow-up, n=5, 5 | -0.024 (0.1638) | -0.014 (0.2812)

43. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocyte MCH for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocyte MCH results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
pg
  Blood erythrocyte MCH, Day 2, n=24, 24, 24 | 0.12 (0.300) | 0.05 (0.292) | 0.05 (0.260)
  Blood erythrocyte MCH, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood erythrocyte MCH, Follow-up, n=3, 2, 3 | 0.03 (0.451) | -0.25 (0.212) | 0.03 (0.252)

44. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocyte MCV for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocyte MCV results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
fL
  Blood erythrocyte MCV, Day 2, n=24, 24, 24 | -0.03 (0.766) | -0.13 (0.761) | 0.29 (0.729)
  Blood erythrocyte MCV, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood erythrocyte MCV, Follow-up, n=3, 2, 3 | 0.07 (1.069) | -0.25 (0.212) | -0.20 (0.100)

45. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils,, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils, Blood Platelets for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils, blood platelets results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles)
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
10^9 cells/Liter
  Blood basophils, Day 2, n=24, 24, 24 | -0.004 (0.0088) | -0.005 (0.0128) | -0.004 (0.0166)
  Blood basophils, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood basophils, Follow-up, n=3, 2, 3 | 0.003 (0.0058) | 0.000 (0.000) | 0.000 (0.0100)
  Blood eosinophils, Day 2, n=24, 24, 24 | -0.028 (0.0478) | -0.024 (0.0460) | -0.019 (0.0482)
  Blood eosinophils, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood eosinophils, Follow-up, n=3, 2, 3 | -0.060 (0.1253) | 0.015 (0.0778) | -0.020 (0.0436)
  Blood leukocytes, Day 2, n=24, 24, 24 | -0.58 (0.925) | -0.75 (1.097) | -0.98 (1.208)
  Blood leukocytes, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood leukocytes, Follow-up, n=3, 2, 3 | -0.63 (1.823) | -2.05 (0.636) | -0.23 (0.643)
  Blood lymphocytes, Day 2, n=24, 24, 24 | -0.057 (0.2571) | -0.105 (0.3268) | -0.196 (0.3254)
  Blood lymphocytes, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood lymphocytes, Follow-up, n=3, 2, 3 | -0.130 (0.5603) | 0.245 (0.2616) | 0.293 (0.2919)
  Blood monocytes, Day 2, n=24, 24, 24 | -0.085 (0.0860) | -0.084 (0.0941) | -0.104 (0.1401)
  Blood monocytes, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood monocytes, Follow-up, n=3, 2, 3 | -0.093 (0.2558) | -0.060 (0.1273) | 0.033 (0.0513)
  Blood neutrophils, Day 2, n=24, 24, 24 | -0.398 (0.8425) | -0.520 (1.0250) | -0.477 (0.8127)
  Blood neutrophils, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood neutrophils, Follow-up, n=3, 2, 3 | -0.350 (0.9560) | -2.225 (0.0919) | -0.563 (0.4179)
  Blood platelets, Day 2, n=24, 24, 24 | 7.4 (15.81) | 12.9 (15.73) | 7.8 (14.96)
  Blood platelets, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood platelets, Follow-up, n=3, 2, 3 | 18.0 (11.14) | 11.0 (29.70) | 12.3 (17.16)

46. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hemoglobin for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood hemoglobin results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles)
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
g/L
  Blood hemoglobin, Day 2, n=24, 24, 24 | 5.0 (5.56) | 6.3 (5.12) | 4.8 (6.65)
  Blood hemoglobin, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood hemoglobin, Follow-up, n=3, 2, 3 | 3.7 (5.69) | 2.0 (5.66) | 3.7 (2.31)

47. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood hematocrit results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles)
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Proportion of red blood cells in blood
  Blood hematocrit, Day 2, n=24, 24, 24 | 0.0126 (0.01745) | 0.0172 (0.01660) | 0.0158 (0.01994)
  Blood hematocrit, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood hematocrit, Follow-up, n=3, 2, 3 | 0.0113 (0.02043) | 0.0090 (0.01697) | 0.0103 (0.00802)

48. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Erythrocytes for Part 2
Description: Blood samples for the assessment of hematology parameters were collected at Baseline and up-to follow-up (Day 36) in Part 2. Baseline was defined as pre-dose assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Data has been presented for blood erythrocytes results for Part 2. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles).
Time Frame: Baseline and up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
10^12 cells/Liter
  Blood erythrocytes, Day 2, n=24, 24, 24 | 0.145 (0.2039) | 0.209 (0.1730) | 0.165 (0.2311)
  Blood erythrocyte, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Blood erythrocyte, Follow-up, n=3, 2, 3 | 0.123 (0.2173) | 0.120 (0.1838) | 0.117 (0.0907)

49. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Method for Part 1
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood and urine protein. In this dipstick test, the level of ketones, glucose, occult blood and protein in urine samples was recorded as negative trace, 1+, 2+, and 3+ (the plus sign increases with a higher level of glucose, ketones, or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up-to follow-up (Day 25) in Part 1. Only categories with significant values have been presented.
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Participants
  Urine Ketones, Trace, Day 2 (-24 hours) | 2 | 2
  Urine Ketones, Trace, Follow-up | 0 | 1
  Urine Occult Blood,Trace,Day 2 (-24 hours) | 0 | 1
  Urine Occult Blood, 1+, Day 2 (-24 hours) | 1 | 0
  Urine Occult Blood, 2+, Day 2 (-24 hours) | 0 | 1
  Urine Occult Blood, 3+, Day 2 (-24 hours) | 1 | 0
  Urine Protein, 3+, Day 2 (-24 hours) | 1 | 0

50. Secondary Outcome: Urine Potential of Hydrogen (pH) Analysis by Dipstick Method for Part 1
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by dipstick method up-to follow-up (Day 25) in Part 1. Only categories with significant values have been presented. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles).
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Points on a scale
  Urine pH, Day 2 (-24 hours), n=14,14 | 6.43 (0.703) | 6.25 (0.672)
  Urine pH, Follow-up, n=5,5: number analyzed (Participants) | 5 | 5
  Urine pH, Follow-up, n=5,5 | 6.20 (0.570) | 6.00 (0.612)

51. Secondary Outcome: Urine Specific Gravity Analysis by Dipstick Method for Part 1
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up-to follow-up (Day 25) in Part 1. Only categories with significant values have been presented. Only those participants with data available at the specified time were analyzed (represented by n=x,x in the category titles).
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Ratio
  Urine Specific Gravity,Day 2(-24 hours),n=14,14 | 1.0131 (0.00871) | 1.0177 (0.00752)
  Urine Specific Gravity,Follow-up,n=5,5: number analyzed (Participants) | 5 | 5
  Urine Specific Gravity,Follow-up,n=5,5 | 1.0180 (0.00831) | 1.0150 (0.01093)

52. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Method for Part 2
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood and urine protein. In this dipstick test, the level of ketones, glucose, occult blood and protein in urine samples was recorded as negative trace, 1+, 2+, and 3+ (the plus sign increases with a higher level of glucose, ketones, or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up-to follow-up (Day 36) in Part 2. Only categories with significant values have been presented.
Time Frame: Up to 36 days in Part 2
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Urine Ketones, Trace, Day 2 (-24 hours) | 1 | 0 | 0
  Urine Occult Blood,Trace,Day 2 (-24 hours) | 1 | 1 | 0
  Urine Occult Blood, 3+, Day 2 (-24 hours) | 1 | 1 | 0
  Urine Occult Blood,1+ Follow-up, | 1 | 0 | 0
  Urine Protein, 1+, Day 2 (-24 hours) | 1 | 0 | 0

53. Secondary Outcome: Urine pH Analysis by Dipstick Method for Part 2
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by dipstick method up-to follow-up (Day 36) in Part 2. Only categories with significant values have been presented. Only those participants with data available at the specified time were analyzed (represented by n=x,x,x in the category titles).
Time Frame: Up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
Number analyzed (Participants) | 24 | 24 | 24
Points on a scale
  Urine pH, Day 2 (-24 hours), n=24, 24, 24 | 6.31 (0.586) | 6.21 (0.641) | 6.31 (0.528)
  Urine pH, Follow-up, n=3, 2, 3: number analyzed (Participants) | 3 | 2 | 3
  Urine pH, Follow-up, n=3, 2, 3 | 5.33 (0.289) | 5.50 (0.000) | 6.83 (0.577)

54. Secondary Outcome: Urine Specific Gravity Analysis by Dipstick Method for Part 2
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up-to follow-up (Day 36) in Part 2. Only categories with significant values have been presented. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Up to 36 days in Part 2
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Treatment C: Participants in this cross-over study received treatment C in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- Treatment D: Participants in this cross-over study received treatment D in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
- Treatment E: Participants in this cross-over study received treatment E in one of the 3 dosing periods in Part 2 as per randomization schedule. The 3 dosing periods were separated by a washout of 7(-4 hours) days between the doses.
Arm/Group | Treatment C | Treatment D | Treatment E
Number analyzed (Participants) | 24 | 24 | 24
Ratio
  Urine Specific Gravity,Day 2(-24 hours),n=24,24,24 | 1.0143 (0.00636) | 1.0148 (0.00515) | 1.0141 (0.00674)
  Urine Specific Gravity,Follow-up,n=3,2,3: number analyzed (Participants) | 3 | 2 | 3
  Urine Specific Gravity,Follow-up,n=3,2,3 | 1.0207 (0.00862) | 1.0165 (0.00354) | 1.0117 (0.00551)

55. Secondary Outcome: Number of Participants With Chemistry Toxicities of Grade 2 as Defined by Division of Acquired Immunodeficiency Syndrome (DAIDS) for Part 1
Description: The DAIDS toxicity table provides descriptive terminology for grading the severity of adult adverse events. Laboratory grades also provide ranges for each parameter. Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: potentially life threatening. low LDL (low-density lipid); HDL (high-density lipid). Data has been presented for clinical chemistry laboratory result parameter (serum sodium) with toxicity of Grade 2 for Part 1.
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Participants | 1 | 0

56. Secondary Outcome: Number of Participants With Urinalysis Toxicities of Grade 2 as Defined by DAIDS for Part 1
Description: The DAIDS toxicity table provides descriptive terminology for grading the severity of adult adverse events. Laboratory grades also provide ranges for each parameter. Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: potentially life threatening, low LDL and HDL Data has been presented for urinalysis laboratory result parameter (urine protein by dipstick analysis) with toxicity of Grade 2 for Part 1.
Time Frame: Up to 25 days in Part 1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg | DTG 50 mg
Number analyzed (Participants) | 14 | 14
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the Day -1 up-to follow-up (25 days for Part 1 and 36 days for Part 2)
Description: All Subjects Population was used for analysis of AEs and SAEs.
Arm/Group | DTG 10 mg | DTG 50 mg | DTG 5 mg (Test 1) | DTG 5 mg (Test 2) | DTG 25 mg (Reference)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14 | 2/24 | 2/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 10 mg (N=14) | DTG 50 mg (N=14) | DTG 5 mg (Test 1) (N=24) | DTG 5 mg (Test 2) (N=24) | DTG 25 mg (Reference) (N=24)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03095638/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT03095638/SAP_001.pdf